CLINICAL TRIAL: NCT00310622
Title: An Assessment of the HyperQ Signal for Detecting Ischemia During Dobutamine Stress Echocardiography (DSE)
Brief Title: Assessment of HyperQ Signal for Detecting Ischemia During Dobutamine Stress ECG
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: BSP Biological Signal Processing Ltd. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SHZ01
Record Dates: First submitted 2006-04-02; First posted 2006-04-04 (Estimated); Last update posted 2007-03-01 (Estimated); Status verified 2007-02

CONDITIONS: Myocardial Ischemia
Keywords: HyperQ; Ischemia; dobutamine
MeSH Terms: conditions — Myocardial Ischemia; Ischemia

INTERVENTIONS:
Device: HyperQ Signal recording

SUMMARY:
The purpose of the study is to verify the ability of the HyperQ signal to detect Dobutamine induced Ischemia. The gold standard for ischemia will be the results of Angiography if performed, or Echocardiographic imaging, which was performed during the test.

DETAILED DESCRIPTION:
Subjects referred for Dobutamine Stress Echocardiography who will sign an Informed consent form will go through the test. High resolution ECG from 12 leads will be recorded using BSP's HyperQ system before, during and following the Echo testing. This wil be done without interfering or affecting any aspect of the normal procedure. Standard Protocol will be used with standard test termination indications.

The Diagnostic stage will include analysis of the hyperQ signal, aiming to classify results as ischemic or non-ischemic.

The HyperQ data will be compared to DSE results which will be used as the "gold standard" for this study unless Angiography results are obtained.

An additional comparison evaluation will be performed to assess the advantage of the HyperQ results on the ST-changes results obtained from conventional ECG.In addition all recruited subjects will be followed for up to 12 months.During this period a phone call will be performed every 3 months to evaluate cardiac status, hospitalization and especially Angiography procedures.

ELIGIBILITY:
Inclusion Criteria:

* Subject referred to dobutamine stress Echocardiography
* Subject signed informed consent

Exclusion Criteria:

* Subjects with implantable Pacemakers or Defibrillators
* Subjects with Wolff-Parkinson-White Syndrome

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150
Dates: Start 2006-03; Study Completion 2007-02

PRIMARY OUTCOMES:
HyperQ Signal recorded during the DES Test

SECONDARY OUTCOMES:
DES Outcome/ Angiography

CONTACTS AND LOCATIONS:
Overall Officials: David Rosenmann, MD, Principal Investigator — Shaarey Zedek Hospital, Jerusalem, Israel
Locations (1):
- Cardiology Department, Shaarey Zedek Hospital, Jerusalem, Israel

REFERENCES:
- See also: Biological Signal Processing Ltd. — http://www.bsp.co.il